CLINICAL TRIAL: NCT03586583
Title: A Feature Comparison Study to Evaluate the Modified Processing of Fujifilm's ASPIRE Cristalle With Digital Breast Tomosynthesis Option as Compared to the Original Processing
Brief Title: Fujifilm Feature Comparison Reader Study to Compare Old vs New Processing
Status: Completed | Type: Observational
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Collaborators: International HealthCare, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: FMSU2017-003
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Results first posted 2020-05-20 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- FBP (old processing): Filtered back projection; old processing.
  Interventions: Device: FBP
- ISR (new processing): Iterative super resolution; new processing.
  Interventions: Device: ISR

INTERVENTIONS:
Device: FBP — Old processing
  Groups: FBP (old processing)
Device: ISR — New processing
  Groups: ISR (new processing)

SUMMARY:
The purpose of the feature comparison study is to evaluate general mammographic features in images of the same breast when reconstructed with modified (ISR and DVIIm) processing as compared to the original processing (FBP with EDR and MFP).

DETAILED DESCRIPTION:
This clinical research is a retrospective, feature comparison reader study with an enriched sample of 600 (100 per radiologist) breast screening or diagnostic cases which were selected from the library of mammograms collected under Fujifilm protocol FMSU2013-004A (all subjects previously provided written informed consent agreeing their image data and supporting documentation could be used for future research and investigations).

Six MQSA-qualified and board-certified mammographers representing various experience levels, will be shown DBT images of a breast with the modified processing side-by-side the same breast with the original processing on the ASPIRE Bellus II workstation.. One breast per subject (two views per breast; CC and MLO) will be evaluated by the readers. Readers will be blinded to the image reconstruction and presentation processing methods. Each reader will be given a different sample of cases to review. Approximately 600 total cases (100 cases per reader) will compose the sample. The order of the subjects and location (left or right review workstation high resolution monitor) of the images with modified processing will be randomized for each reader.

The primary objective is the readers' assessment for each of the 7 general mammographic features. The null hypothesis is that the pooled proportion of cases judged as non-inferior with modified image processing is <0.50, versus the alternative hypothesis that the pooled proportion is >0.50. If the 95% CI does not contain values <0.50, then the null hypothesis will be rejected. These hypotheses will be evaluated for each of the 7 general mammographic features. If all 7 null hypotheses are rejected, then it will be concluded that the modified imaging features are non-inferior to the original imaging

ELIGIBILITY:
Inclusion Criteria:

* Female subjects participating in FMSU2013-004A protocol with known clinical status

Exclusion Criteria:

* Female subjects that did not have known clinical status in FMSU2013-004A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 600
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Crennan, Study Director — Fujifilm Medical Systems USA, Inc.
Locations (1):
- International HealthCare, LLC, Norwalk, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 qualified radiologists were shown DBT (Tomosynthesis) of a breast with the modified processing side-by-side the same breast with the original processing. Each reader was given a unique sample of 100 cases to review. Images were acquired under Fujifilm image acquisition protocol FMSU2013-004A
Groups:
- FBP (Old Processing) and ISR (New Processing): Radiologists reviewed images of a breast with ISR side-by-side the same breast with FBP. They were blinded to the image reconstruction and presentation processing methods. Radiologists compared several general mammographic features and were asked to grade each feature on each view using the 5-point Likert scale outlined previously.
Period: Overall Study
Arm/Group | FBP (Old Processing) and ISR (New Processing)
Started | 600
Completed | 600
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- FBP (Old Processing)/ISR (New Processing): Filtered back projection (old processing) and ISR (new processing) images of the same breast are presented side-by-side for radiologist review.
Arm/Group | FBP (Old Processing)/ISR (New Processing)
Number analyzed (Participants) | 600
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 563
  >=65 years | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 600
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 590
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 600

OUTCOME MEASURES:

1. Primary Outcome: Comparison of ISR (Modified Processing) to FBP (Original Processing)
Description: For each reader, the cases judged as non-inferior with modified processing will be calculated for each feature and each view. Non-inferiority will be defined as a score of equivalence between modified and original or a score indicating the modified image processing is superior. Readers compared several general mammographic features using the following 5-point scale:
  negative 2 (left image much superior) negative 1 (left image somewhat superior) 0 (left and right images are equivalent) positive 1 (right image somewhat superior) positive 2 (right image much superior)
Time Frame: 1 day reading session
Population: Six readers read a cohort of images acquired under a prior acquisition study protocol (FMSU2013-004A). Statistician provided results for ISR (modified/new processing only) that was already analyzed/compared to FBP (old processing).
Measure: Mean (95% Confidence Interval); unit: 5-point scale
Arm/Group | ISR (New Processing)
Number analyzed (Participants) | 600
5-point scale
  MLO | 0.83 [0.66 to 0.95]
  Uniformity | 0.83 [0.68 to 0.95]
  Contrast | 0.80 [0.66 to 0.90]
  Sharp | 0.79 [0.67 to 0.89]
  Skin | 0.84 [0.68 to 0.96]
  Noise | 0.83 [0.69 to 0.95]
  Artifact | 0.84 [0.69 to 0.95]
  Mass | 0.63 [0.49 to 0.75]
  Calcification | 0.87 [0.78 to 0.94]
  Arch Distortion/Asymmetry | 0.64 [0.45 to 0.79]

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: There were no AE's expected for this study, as it was a radiologist reader study utilizing retrospective imaging. No study subjects were on-site for this retrospective review. No Adverse Events to report.
Groups:
- FBP (Old Processing); ISR (New Processing): This was a reader study where radiologists/readers compared processing of previously acquired images.
Arm/Group | FBP (Old Processing) | ISR (New Processing)
All-Cause Mortality (participants affected / at risk) | 0/600 | 0/600
Serious Adverse Events (participants affected / at risk) | 0/600 | 0/600
Other Adverse Events (participants affected / at risk) | 0/600 | 0/600

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT03586583/Prot_003.pdf
  • Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT03586583/SAP_002.pdf